CLINICAL TRIAL: NCT00753220
Title: A Phase I/IIa Trial of Combined Cryotherapy and Intra-tumoral Immunotherapy With Autologous Immature Dendritic Cells (VDC2008) in Chemo-naïve Men With Prostatic Adenocarcinoma and Limited Metastases to Lymph Nodes and/or Bone
Brief Title: Safety Study of Autologous Dendritic Cells Injected Into the Prostate After Cryoablation for Advanced Prostate Cancer
Acronym: CRITICAL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrew the IND with the FDA.
Sponsor: Bostwick Laboratories (Industry)
Collaborators: Prostate Institute of America (Unknown); Community Memorial HealthCenter (Other); HemaCare Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRITICAL001
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Androgen; Independent; Prostate Cancer; (AIPC),; Hormone-refractory; (HRPC),; cryotherapy,; dendritic cell,; immunotherapy; Chemo-naïve; lymph nodes; bone
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VDC2008 (Experimental): Cryoablation of prostate followed by dendritic cell injection (dose of 2.5 x 10^7, 7.5 x 10^7, or 1.0 x 10^8 cells depending on assigned cohort) into prostate and low dose cyclophosphamide therapy (dose: 25 mg, p.o., b.i.d. for 7 days on and 7 days off; a total of 6 cycles [1 cycle = 4 weeks] starting Week 2 after cryoablation and going to Week 26)
  Interventions: Biological: VDC2008; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: VDC2008 — Intratumoral injection of VDC2008 post-cryotherapy.
  Dosage will depend on cohort: 2.5 x 10^7, 7.5 x 10^7 or 1.0 x 10^8 cells
  Other Names: Autologous dendritic cells
Drug: Cyclophosphamide — Cyclophosphamide i.v. given at day -3 (dose: 300mg/m2); Low-dose Cyclophosphamide pill given twice daily (dose: 25 mg, p.o., b.i.d. for 7 days on and 7 days off; a total of 6 cycles [1 cycle = 4 weeks] starting Week 2 after cryoablation and going to Week 26)

SUMMARY:
The purpose of this study is to determine if the intra-tumoral injection of a subject's own dendritic cells after cryotherapy of the prostate is a safe and effective treatment for advanced prostate cancer.

In theory, the injected dendritic cells will internalize antigens from the tumor cells which have been damaged by cryotherapy and activate the subject's immune system against that specific tumor.

Subjects will also receive a low dose chemotherapy designed to lower the number of T-regulatory cells which have been shown to lower or stop some immune system responses.

Hypothesis 1: Dendritic cell injection into cryotreated prostate cancer is non-toxic;

Hypothesis 2: Dendritic cell injection into cryotreated prostate cancer is medically beneficial to the subject.

DETAILED DESCRIPTION:
The study treatment dendritic cells (VDC2008) will be injected into the prostate following prostatic cryoablation. It is speculated that antigen from the cryoablated cancer will be available in the vicinity of the cryoablation field immediately following the procedure. Autologous, immature dendritic cells are capable of internalizing antigen, migrating to the lymphatic system, and presenting antigenic epitopes to T lymphocytes. In this way, dendritic cells are capable of initiating a cell-mediated systemic immune response.

In concept, the cancer itself should provide a specific and potentially broad spectrum of cancer-related antigens. Regulatory T lymphocytes, which have been implicated in dampening or halting cell-mediated, antigen-specific immune responses, will be selectively depleted using a regimen of low-dose cyclophosphamide. Low-dose cyclophosphamide has been empirically shown to selectively deplete the number of circulating regulatory T cells.

Using this combination of therapies, it is thought that a clinically significant anti-cancer immune response might be elicited.

ELIGIBILITY:
Inclusion Criteria

* Men ≥ 18 years of age and any race.
* Signed Informed Consent document obtained prior to the initiation of screening procedures.
* Histologically documented primary adenocarcinoma of the prostate. A specimen of the primary tumor must be submitted to the Central Pathology Laboratory for confirmation of prostatic adenocarcinoma and determination of Gleason Sum grading.
* Prior history of:

  1. Androgen Deprivation Therapy; or
  2. Organ-preserving therapy (i.e., non-prostatectomy) for primary prostate cancer (e.g., radiation therapy).
* In case of recurrence, subject must have evidence of prostate cancer by a positive biopsy revealing adenocarcinoma within the past 6 months of screening and confirmed by the Central Pathology Laboratory.
* TxNxM1a and/or TxNxM1b disease limited to three total metastatic sites as evidenced by lymph node metastases and /or bone metastases at time of screening.

  1. TxNxM1a : Lymph node metastases histologically proven and confirmed by Central Pathology Laboratory;
  2. TxNxM1a: Lymph node metastases not histologically proven, given that the following are satisfied in the temporal order listed:

     1. Computed tomography (CT) or Magnetic Resonance Imaging (MRI) for positive lymph nodes negative at original diagnosis of prostate cancer;
     2. Definitive local treatment undertaken;
     3. Evidence of local treatment failure on the basis of rising serum PSA;
     4. Prostatic biopsy positive for carcinoma;
     5. Subsequent CT or MRI reveals lymph node(s) of 2 cm diameter or greater
  3. TxNxM1b: Bone metastases demonstrated by radionuclide bone scan, CT, or MRI.
* Androgen-independent prostate cancer as defined by:

  1. Three consecutive rises of at least 10% each in serum PSA, in which all serum PSA measurements are separated by at least one week and results are obtained within 60 days of study screening; OR
  2. Three rises that involve an increase of 50% over the nadir serum PSA, in which all serum PSA measurements are separated by at least one week and results are obtained within 60 days of study screening;
  3. A castrate level of testosterone (<50 ng/dl) obtained within 60 days of study screening.
* Life expectancy of greater than or equal to 12 months.
* Adequate hematological function as defined by:

  1. Total WBC > 4,500/mm3
  2. Total lymphocyte count > 500/mm3
  3. Hemoglobin > 12.0 g/dl
  4. Neutrophils > 1,500/mm3
  5. Platelets > 150,000/mm3
* Adequate renal function with creatinine < 2.0 mg/dl.
* Adequate liver function as defined by:

  1. AST and ALT < 2 times the upper limit of normal;
  2. Serum bilirubin < 2.0 mg/dl;
  3. Alkaline Phosphatase < 2.0 upper limit of normal.
* Assessment of superficial veins as adequate for the performance of leukapheresis.
* No active major medical or psychological problems that could be complicated by study participation.

Exclusion Criteria

* The presence of lung, liver or brain metastases, malignant pleural effusions or malignant ascites.
* Moderate or severe symptomatic metastatic disease. Subjects who meet either of the following criteria must be excluded:

  1. A requirement for treatment with opioid analgesics for any reason within 21 days prior to study screening;
  2. Average weekly pain score of 4 or more as reported on the 11-point Pain Intensity - Numerical Rating Scale (Appendix III) over the two weeks prior to study enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2 accessed at study screening visit.
* Chemotherapy treatment at any time prior to study screening.
* Radiation therapy for metastatic disease, including intravenous radioactive strontium therapy.
* Initiation or discontinuation of bisphosphonate therapy within 28 days prior to study screening. Subjects taking bisphosphonate medication must not have their dosing regimen altered until objective disease progression is independently confirmed.
* Treatment with any of the following medications or interventions within 28 days of study screening:

  1. Systemic corticosteroids (use of inhaled, intranasal and topical steroids is acceptable);
  2. External beam radiation therapy or surgery;
  3. PC-SPES (or PC-SPEC) or Saw Palmetto extract;
  4. Megestrol acetate (Megace®), diethyl stilbesterol (DES), or cyproterone acetate;
  5. Ketoconazole;
  6. High dose calcitriol (i.e., > 7.0 μg/week);
  7. Any other systemic therapy for prostate cancer.
* Treatment with any investigational vaccine within 2 years of enrollment to this study.
* Treatment with any other investigational product within 28 days of study screening.
* Pathologic long-bone fractures, imminent pathologic long-bone fracture (cortical erosion on radiography > 50%) or spinal cord compression.
* Impending untreated spinal cord compression or urinary outlet obstruction.
* Paget's Disease of bone.
* History of stage III or greater cancer, excluding prostate cancer:

  1. Basal or squamous cell skin cancers must have been adequately treated and the subject must be disease-free at the time of study screening visit;
  2. Subjects with a history of stage I or II cancer must have been adequately treated and be disease-free for ≥ 3 years at the time of study screening
* Requirement for systemic immunosuppressive therapy for any reason
* Prior or currently active autoimmune disease requiring management with systemic immunosuppression. Such conditions include inflammatory bowel disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-related thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatological disease.
* Any infection requiring parenteral antibiotic therapy or causing fever (body temperature > 100.5°F or 38.1°C) within 1 week prior to study screening.
* Known allergy, intolerance, or medical contraindication to receiving the contrast dye required for the protocol-specified CT imaging
* History of asthma, anaphylaxis, or other known serious adverse reactions to vaccines.
* Any medical intervention or other condition which, in the opinion of the Physician-Investigator could compromise adherence with study requirements or otherwise compromise study subject safety and the study's objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duke K Bahn, M.D., Principal Investigator — Prostate Institue of America
Locations (1):
- Community Memorial Hospital, Ventura, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men at least 18 years of age diagnosed with prostate cancer with metastases limited to three sites (e.g., lymph nodes and/or bone) who have been determined to have undergone progression of their cancer under androgen blockade (i.e., are androgen-independent) will be eligible for this study.
Pre-assignment Details: Prior to any screening evaluations, the purpose of the study & study related tests/procedures will be explained, then subject signs ICF. Subject will undergo screening assessments to determine if he meets all of the inclusion criteria & none of the exclusion criteria. Screen failures will not be eligible for re-screening.
Groups:
- VDC2008: Cryoablation of prostate followed by dendritic cell injection into prostate and low dose cyclophosphamide therapy
  VDC2008 : Intratumoral injection of VDC2008 post-cryotherapy.
  Dosage will depend on cohort: 2.5 x 10^7, 7.5 x 10^7 or 1.0 x 10^8
Period: Overall Study
Arm/Group | VDC2008
Started | 7
Completed | 2
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | VDC2008
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: PROTOCOL EXCERPT: The primary objective of the Phase I Portion of this study is the determination of the maximum tolerated dose (MTD) of intratumorally injected study agent VDC2008 administered following cryoablation of the prostate, and pre- and post-treatment with a low-dose cyclophosphamide therapy, as determined by toxicity and adverse event monitoring following treatment of metastatic androgen-independent prostate cancer.
  ADDITIONAL INFORMATION: MTD was not reached by any study participant prior to end of the study. Additional participants would have been necessary to determine MTD.
Time Frame: Up to 1 year
Measure: Number; unit: intratumorally delivered cells
Arm/Group | VDC2008
Number analyzed (Participants) | 7
intratumorally delivered cells | NA — MTD was not reached by any study participant prior to end of the study.

ADVERSE EVENTS:
Time Frame: Overall Study (1 year, 2 months)
Arm/Group | VDC2008
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VDC2008 (N=7)
Memory (Nervous system disorders) | 1 (1) — Memory Problem from General Anesthesia
Heartburn (Gastrointestinal disorders) | 1 (1) — Mild heartburn
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Loss of Appetite (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No